CLINICAL TRIAL: NCT01050179
Title: Chemoreflex Gain on Exercise
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Darrel Francis, Imperial College
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10/H0712/9
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Last update posted 2010-04-19 (Estimated); Status verified 2010-04

CONDITIONS: Exertional Periodic Breathing
Keywords: chemosensitivity
MeSH Terms: interventions — Carbon Dioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: carbon dioxide — sinusoidal carbon dioxide delivery

SUMMARY:
The purpose of this study is to assess chemoreflex gain on exercise.

DETAILED DESCRIPTION:
Normally breathing is controlled by a reflex that responds to the levels of carbon dioxide (CO2) in the blood. The change in breathing that results from a change in the blood's CO2 concentration is called the chemoreflex.

In heart failure, a condition where the heart muscle is damaged and can not pump as well, this reflex is exaggerated. The result of this can be breathing conditions characterised by patients hyperventilating at times and at other times taking very shallow breaths or even stopping altogether. In the past the only way of measuring this chemoreflex was to get patients to breathe into a large container and to rebreathe their exhaled air and allow the CO2 to rise over time, whilst keeping the oxygen constant. The proportion by which the ventilation increases with increasing carbon dioxide is the chemoreflex gain. Unfortunately, because this test takes a long time to conduct, requires specialist knowledge and equipment it has not been possible to measure this reflex on exercise.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers: Males aged 18-80 years who are able to perform both running and cycling and can follow simple visual instructions.
* Heart Failure Subjects: Males aged 18-80 with a clinical diagnosis of heart failure who are able to perform both running and cycling and can follow simple visual instructions.

Exclusion Criteria:

* Chest pain of any cause within 4-6 days,
* Pulmonary oedema,
* Uncontrolled hypertension (systolic blood pressure > 220 mm Hg, diastolic >120 mm Hg),
* Severe aortic stenosis,
* Severe hypertrophic obstructive cardiomyopathy,
* Untreated life threatening arrhythmia,
* Dissecting aneurysm,
* Recent surgery (within 4-6 weeks), COPD.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
chemoreflex gain on exercise | every minute

SECONDARY OUTCOMES:
Reproducibility of chemoreflex gain on exercise | every minute

CONTACTS AND LOCATIONS:
Locations (1):
- St Mary's Hospital, Paddington, London, United Kingdom